CLINICAL TRIAL: NCT05390255
Title: Establishment of Precise Diagnosis and Treatment System for Refractory Chronic Rhinosinusitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TR-system for RCRS
Record Dates: First submitted 2022-05-06; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Sinusitis
Keywords: Refractory chronic sinusitis; Randomized Controlled Trial; Hormone therapy; Omalizumab; Biomarkers
MeSH Terms: conditions — Sinusitis | interventions — Hormones; Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nasal spray hormone therapy (Experimental): This group of patients received nasal steroid therapy throughout the study. The clinical data of patients at baseline and each visit period were collected, the incidence of adverse events was recorded, and the short-term efficacy and safety of different drug treatment regimens were evaluated.
  Interventions: Drug: Mometasone furoate nasal spray hormone
- Nasal spray hormone therapy + oral hormone therapy (Experimental): The patients in this group were given oral hormone therapy for 14 days in the first month and the fourth month under the background of nasal spray hormone treatment throughout the course. The clinical data of patients at baseline and each visit period were collected, the incidence of adverse events was recorded, and the short-term efficacy and safety of different drug treatment regimens were evaluated.
  Interventions: Drug: Mometasone furoate nasal spray hormone + oral hormone
- Nasal spray hormone therapy + omalizumab therapy (Experimental): The patients in this group were injected with omalizumab once a month under the background of nasal spray hormone therapy, for a total of 6 times. The clinical data of patients at baseline and each visit period were collected, the incidence of adverse events was recorded, and the short-term efficacy and safety of different drug treatment regimens were evaluated.
  Interventions: Drug: Mometasone furoate nasal spray hormone + omalizumab

INTERVENTIONS:
Drug: Mometasone furoate nasal spray hormone — This group of patients received mometasone furoate nasal spray hormone treatment throughout the study.
  Arms: Nasal spray hormone therapy
Drug: Mometasone furoate nasal spray hormone + oral hormone — The patients in this group were given oral hormone therapy for 14 days in the first month and the fourth month under the background of mometasone furoate nasal spray hormone treatment throughout the course.
  Arms: Nasal spray hormone therapy + oral hormone therapy
Drug: Mometasone furoate nasal spray hormone + omalizumab — The patients in this group were injected with omalizumab once a month under the background of mometasone furoate nasal spray hormone treatment, for a total of 6 times.
  Arms: Nasal spray hormone therapy + omalizumab therapy

SUMMARY:
Chronic rhinosinusitis that recurs after adequate surgery and conventional medical treatment is called refractory chronic rhinosinusitis (RCRS). Omalizumab and oral glucocorticoid therapy can play an important role in the treatment of RCRS, but there is still a lack of comparative studies on the efficacy and safety of the two. In addition, biomarkers are a hotspot in RCRS research, but there is still a lack of studies on changes in marker expression with disease progression and treatment.

In this study, patients aged 18-70 who were diagnosed with CRS were consecutively enrolled, and the patients were divided into RCRS and non-RCRS groups according to pathological results. The patients in the RCRS group were randomly divided (1:1:1) into the nasal spray hormone therapy group, the nasal spray hormone therapy + oral hormone therapy group, and the nasal spray hormone therapy + omalizumab therapy group by a multi-center, randomized, controlled study. The patients were treated for 6 months and followed up for 6 months after treatment. Clinical data such as symptom score and endoscopic score before and after treatment were collected, adverse events were recorded, and the differences in efficacy and safety among the groups were compared. Non-invasive samples such as nasal secretions and exfoliated cells were collected, and the expression and variation of different immune intrinsic markers were explored combined with follow-up results. The development of this project contributes to the establishment of a precise diagnosis and treatment system for refractory chronic sinusitis.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18-70 years old;
* (2) All meet the diagnostic criteria of CRS in EPOS2020;
* (3) Patients with asthma were in a stable state, with FEV1 > 80% of the predicted value or 80% of the optimal value of personal FEV1;
* (4) Good compliance, able to complete clinical observation. Meet the diagnostic criteria for RCRS that the number of eosinophils per high power field in the nasal mucosa is >55 or the percentage of eosinophils in the tissue is ≥27%;
* (5) Investigator-assessed endoscopic bilateral Nasal Polyp Size Score (NPSS) of 4-6 (minimum score of 2 per nasal cavity);
* (6) Male or eligible female subjects (female subjects not pregnant or breastfeeding);
* (7) Ability to sign an informed consent form, including compliance with the requirements and restrictions outlined in the Informed Consent Form (ICF) and this protocol.

Exclusion Criteria:

* (1) Medication history of oral glucocorticoids within 3 months before enrollment, glucocorticoid atomization treatment and nasal hormone spray treatment within 2 weeks;
* (2) Oral glucocorticoid contraindications, such as diabetes, femoral head necrosis, gastric ulcer, etc.;
* (3) Any nasal and/or sinus surgery within 3 months before enrollment;
* (4) Patients have conditions or comorbidities that may preclude evaluation of the primary efficacy endpoint, such as: unilateral posterior nasal polyp of maxillary sinus, acute rhinitis, nasal infection or upper respiratory tract at the screening period or within 2 weeks before the screening period infection, acute asthma attack within 4 weeks, current drug-induced rhinitis, allergic fungal sinusitis (AFRS), benign or malignant tumor of nasal cavity, severe nasal septal deviation (Obstruction of one nostril, preventing full evaluation of nasal polyps in both nostrils), undergoing sinus or sinus surgery to alter the structure of the nasal wall resulting in an inability to evaluate the nasal polyp score, persistent drug-induced rhinitis (rebound or chemical-induced rhinitis);
* (5) Important clinical comorbidities that may interfere with clinical effectiveness, including but not limited to: active upper or lower respiratory tract infection, cystic fibrosis, eosinophilic granuloma with polyvasculitis (Churg-Strauss syndrome), granulomatosis with polyangiitis (Wegener's granulomatosis), Young's syndrome, etc.;
* (6) Accompanying serious diseases or recurrent chronic diseases with poor systemic control, such as (but not limited to), active infection, cardiovascular disease, tuberculosis or other pathogen infection, diabetes, autoimmune disease, HIV, hepatitis B, Hepatitis C or parasitic diseases, malignant tumors, etc.;
* (7) Subjects with severe liver and kidney function injury; such as, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >2 times the upper limit of normal, serum creatinine > the upper limit of normal value; liver cirrhosis or currently unstable liver or biliary disease as assessed by the investigator;
* (8) Known or suspected immunosuppression, including a history of invasive opportunistic infections (such as tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pulmonary cysts, aspergillosis), even if the infection has subsided;
* (9) Suffering from known, pre-existing, clinically significant cardiac, endocrine, autoimmune, metabolic, neurological, renal, hepatic, hematological or other systemic abnormalities that have not been controlled by standard treatment;
* (10) Patient has been exposed to ionizing radiation above background 10mSv in the past 3 years due to occupational exposure or previous study participation (excluding clinically reasonable therapeutic or diagnostic exposure);
* (11) Women who were pregnant or planned to become pregnant during the study, or who were breastfeeding;
* (12) Subjects who were fertile but were reluctant to use medically approved and effective contraception;
* (13) Those with a history of alcohol or drug abuse;
* (14) Those who had been treated with monoclonal antibodies in the 6 months prior to enrollment;
* (15) Those who believed the patient had other medical or non-medical conditions that were not suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in endoscopic score | Baseline, week 2, week 4, week 8, week 12, week 14, week 16, week 20, week 24, month 9, month 12
  Bilateral polyp volume size described using the Nasal Polyp Size Score (NPSS) score. (0 - 4 points per side: 0 = no polyp; 1 = small polyp in the middle meatus, not reaching the inferior border of the middle turbinate; 2 = small polyp in the middle meatus, reaching the inferior border of the middle turbinate; 3 = large polyp protruding from the middle meatus, not reaching the inferior border of the inferior turbinate; 4 = large polyp that almost causes most or complete obstruction of the nasal cavity.)

SECONDARY OUTCOMES:
The change in nasal symptoms | Baseline, week 2, week 4, week 8, week 12, week 14, week 16, week 20, week 24, month 7, month 8, month 9, month 10, month 11,month 12
  Nasal symptom was assessed using the Visual Analog Scale (VAS). The symptoms are graded on a 10-point scale (0 = no symptoms; 10 = most severe symptoms).
The change in sinus CT score | Baseline, week 24
  The Lund-Mackay imaging scoring system was used for the CT scan results of the sinuses (0, 1, and 2 were used for each frontal sinus, anterior ethmoid sinus, posterior ethmoid sinus, maxillary sinus, and sphenoid sinus, indicating no opacity, partial opacity and all turbidity of the sinus cavity respectively; 0 and 2 were used for each side of the sinus complex to indicate no blockage and presence of blockage) to calculate the total score and E/M value (bilateral ethmoid total score/bilateral maxillary sinus total score), etc.
The change in SNOT-22 score | Baseline, week 2, week 4, week 8, week 12, week 14, week 16, week 20, week 24, month 7, month 8, month 9, month 10, month 11,month 12
  The 22-item Sino-nasal outcome test (SNOT-22) was used to evaluate the changes in symptoms of patients. According to the severity of symptoms caused by RCRS, each item was divided into 6 levels: no distress (0 points), mild distress (1 point), mild distress (2 points) ), moderate distress (3 points), severe distress (4 points), very severe distress (5 points). The higher the score, the more severe the symptoms, and the final total score of the item is counted.
The change in exfoliated cells and secretions | Baseline, week 2, week 4, week 8, week 12, week 14, week 16, week 20, week 24, month 9,month 12
  Changes in expression levels of T1, T2, T3 factors and T2 inflammatory markers CST1 and CLC in nasal brush exfoliated cells and nasal secretions.
The change in asthma ACQ Score | Baseline, week 2, week 4, week 8, week 12, week 14, week 16, week 20, week 24, month7, month 8, month 9, month 10, month 11, month 12
  For patients with asthma, we assessed the change of asthma symptoms through the Asthma Control Questionnaire (ACQ). Each question was scored on a scale of 0 to 6 according to the severity. The result score of each item was averaged. A score of <0.75 indicated that the asthma had been completely controlled; a score of 0.75-1.5 indicates well-controlled asthma; a score of >1.5 indicates that asthma is not controlled.
The change in AE / SA recording | Baseline, week 2, week 4, week 8, week 12, week 14, week 16, week 20, week 24, month7, month8, month 9, month 10, month 11, month 12
The change in serum cortisol | Baseline, week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No